CLINICAL TRIAL: NCT02469298
Title: A Randomized, Double-blind, Placebo Controlled Study to Evaluate the Safety, Tolerability and Clinical Effect of Oral Danirixin (GSK1325756) in the Treatment of Healthy Adults With Acute, Uncomplicated Influenza (201682)
Brief Title: Safety, Tolerability and Clinical Effect of Danirixin in Adults With Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201682
Record Dates: First submitted 2015-04-23; First posted 2015-06-11 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Virus Diseases
Keywords: acute, uncomplicated influenza; Danirixin; oseltamivir
MeSH Terms: conditions — Virus Diseases | interventions — danirixin; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Danirixin + Oseltamivir matching placebo (Experimental): Subjects will receive 75 mg oral Danirixin twice daily with Oseltamivir matching placebo twice daily for a total of ten doses over five days
  Interventions: Drug: GSK1325756 (Danirixin); Drug: Placebo To Match Oseltamivir Phosphate
- Danirixin matching placebo + Oseltamivir matching placebo (Placebo Comparator): Subjects will receive Danirixin matching placebo twice daily with Oseltamivir matching placebo twice daily for a total of ten doses over five days
  Interventions: Drug: Placebo To Match GSK1325756; Drug: Placebo To Match Oseltamivir Phosphate
- Danirixin + Oseltamivir (Experimental): Subjects will receive 75 mg oral Danirixin twice daily with 75 mg Oseltamivir twice daily for a total of ten doses over five days
  Interventions: Drug: GSK1325756 (Danirixin); Drug: Oseltamivir Phosphate
- Danirixin matching placebo + Oseltamivir (Active Comparator): Subjects will receive Danirixin matching placebo twice daily with 75 mg Oseltamivir twice daily for a total of ten doses over five days
  Interventions: Drug: Placebo To Match GSK1325756; Drug: Oseltamivir Phosphate

INTERVENTIONS:
Drug: GSK1325756 (Danirixin) — It will be supplied as capsule shaped white film coated tablet containing 75 mg GSK1325756 for oral use
  Arms: Danirixin + Oseltamivir; Danirixin + Oseltamivir matching placebo
Drug: Placebo To Match GSK1325756 — It will be supplied as capsule shaped white film coated placebo tablet for oral use
  Arms: Danirixin matching placebo + Oseltamivir; Danirixin matching placebo + Oseltamivir matching placebo
Drug: Oseltamivir Phosphate — It will be supplied as size 0 Swedish Orange capsule containing 75 mg Oseltamivir phosphate and overfill of pre-gelatinized starch for oral use
  Arms: Danirixin + Oseltamivir; Danirixin matching placebo + Oseltamivir
Drug: Placebo To Match Oseltamivir Phosphate — It will be supplied as size 0 Swedish Orange capsule containing pre-gelatinized starch and magnesium stearate for oral use
  Arms: Danirixin + Oseltamivir matching placebo; Danirixin matching placebo + Oseltamivir matching placebo

SUMMARY:
Study 201682 is a Phase IIa, randomized, double blind, placebo-controlled four arm outpatient study evaluating the safety, tolerability and clinical effect of danirixin or danirixin + oseltamivir combination in comparison to placebo or oseltamivir twice daily for 5 days in otherwise healthy adults with laboratory confirmed influenza infection. Danirixin is a selective and reversible C-X-C Chemokine Receptor 2 (CXCR2) antagonist that inhibits neutrophil transmigration and activation to areas of inflammation. The study endpoints are intended to test the hypothesis that inhibition of neutrophil activation by approximately 50-60% (as previously measured by cluster of differentiation [CD11b] expression in response to chemokine [C-X-C motif] ligand 1 [CXCL1] stimulation ex vivo in human studies) will not impact safety parameters or worsen clinical manifestations of disease, disease-related events of interest, or viral load, and may possibly improve these parameters when administered within 48 hours of symptom onset. The aim of this exploratory study is to obtain data on the safety, tolerability and clinical effect of GSK1325756 (danirixin [DNX]) alone or in combination with oseltamivir (OSV) in otherwise healthy adults with acute, uncomplicated influenza prior to future evaluation in hospitalized patients with complicated influenza. The primary objective is to assess safety and tolerability of DNX with and without a neuraminidase inhibitor through the evaluation of AEs, SAEs, clinical laboratory tests, vital signs, and electrocardiogram (ECG) parameters. Safety assessments will also include an assessment of disease related events (DREs) of interest and associated antibiotic use. The Influenza Intensity and Impact Questionnaire (FluiiQ™) will be used in the study to document patient reported outcomes (PROs). The screening visit in Australia will be composed of a pre-screen for influenza infection with an influenza rapid antigen test followed by a screen for the remaining eligibility criteria for those subjects with a positive result on the influenza rapid antigen test. FluiiQ is trademark owned by Measured Solutions for Health Private Limited.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 64 years of age inclusive, at the time of signing the informed consent;
* Onset of influenza-like illness symptoms within 48 hours prior to study enrollment. Onset of symptoms is defined as the time when the subject's temperature was measured as elevated (>=38.0°C [>=100.4°F]) OR the time when the subject first experienced at least one symptom (cough, sore throat, nasal congestion, headache, feeling feverish, body aches and pains, or fatigue);
* Subjects have an oral temperature >=38.0°C (>=100.4°F) at screening visit or history of feeling feverish within the 24 hours prior to screening visit;
* At least one respiratory symptom (cough, sore throat, nasal congestion) and at least one systemic symptom (headache, body aches and pain, fatigue) due to influenza infection;
* A positive influenza rapid antigen test;
* Body weight >60 Kilogram (kg) for men and >45 kg for women; and Body Mass Index (BMI) between 19 to 35 kilogram per meters squared (kg/m^2), inclusive;
* Male or Female subjects could be eligible if :

Male subjects with female partners of child-bearing potential must comply with the following contraception requirements from the time of first dose of study medication until at least 36 hours (five half-lives) of study medication after the last dose of study medication:

Vasectomy with documentation of azoospermia; Male condom plus partner use of one of the following contraceptive options: Contraceptive subdermal implant; Intrauterine device or intrauterine system; Oral Contraceptive, either combined or progestogen alone; Injectable progestogen; Contraceptive vaginal ring ; Percutaneous contraceptive patches; This is an all-inclusive list of those methods that meet the following GlaxoSmithKline (GSK) definition of highly effective: having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. For non-product methods (e.g., male sterility), the investigator determines what is consistent and correct use. The GSK definition is based on the definition provided by the International Conference on Harmonisation (ICH). The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception;

* Female subject: is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies

Non-reproductive potential defined as:

Pre-menopausal females with one of the following: documented Tubal ligation; Documented Hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study.

Reproductive potential agrees to follow one of the options listed below in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from the time of screening, during dosing, and until at least 36 hrs after the last dose of study medication and completion of the follow-up visit.

GSK List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) meeting GSK criteria of highly effective: having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penilevaginal intercourse on a long term and persistent basis.

Contraceptive subdermal implant; Intrauterine device or intrauterine system; Combined estrogen and progestogen oral contraceptive; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

- Subjects willing and able to give written informed consent to participate in the study and to adhere to the procedures stated in the protocol.

Exclusion Criteria:

- Subject defined as being at high risk of complications from influenza infection according to the World Health Organization (WHO) Guidelines for Pharmacological Management of Pandemic Influenza A (H1N1) and other Influenza Viruses: Pregnant women; Persons of any age with chronic pulmonary disease (e.g. Mild persistent, Moderate or severe asthma, Chronic Obstruction Pulmonary Disease [COPD], cystic fibrosis, bronchiectasis); Persons of any age with chronic cardiac disease (e.g. congestive cardiac failure);

* Persons with metabolic disorders (e.g. diabetes); Persons with chronic renal disease, chronic hepatic disease, certain neurological conditions (including neuromuscular, neurocognitive and seizure disorders, but not including autism spectrum disorders); Hemoglobinopathies, or immunosuppression, whether due to primary immunosuppressive conditions, such as Human Immunodeficiency Virus (HIV) infection, or secondary conditions, such as immunosuppressive medication or malignancy;
* Subjects in whom treatment with an influenza antiviral is considered essential;
* Severity of illness requiring or anticipated to require in-hospital care;
* Pulse Oximetry levels <92% (at rest on room air) at screening or requirement for supplemental oxygen;
* Any complication of respiratory tract infection, signs of severe or progressive disease, or worsening of any pre-existing medical condition at the time of enrollment, that, in the opinion of the investigator, would place the subject at an unreasonably increased risk of participation in this study;
* Suspicion or confirmation of bacterial infection (e.g. otitis media, sinusitis, bronchitis, focal pneumonia) or who are requiring oral or systemic antibiotics within one week before enrollment;
* Women who are pregnant as determined by a positive urine human chorionic gonadotrophin (hCG) test prior to dosing or women who are breastfeeding;
* Current or chronic documented history of liver disease (including Hepatitis A, B, or C), or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones); In this case "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records). In questionable cases the subject cannot be enrolled;
* Corrected QT interval (QTc) >450 millisecond (msec) or QTc >480 msec in subjects with Bundle Branch Block.
* Subjects currently using or expected to use: oral or injectable Cytochrome P450 3A4 (CYP3A4) or Breast Cancer Resistance Protein (BCRP) substrates with a narrow therapeutic index, or oral or systemic glucocorticoids during the study period; Antacids can be used but should not be taken for at least 3 hours preceding and 2 hours after administration of study drug; proton pump inhibitors and histamine H2-receptor antagonists are prohibited from the screening visit until 12 hours after completion of the final dose of study treatment.
* Subjects who have taken an approved or investigational anti-influenza medication (e.g., oseltamivir, zanamivir, peramivir, laninamivir, amantadine, rimantidine, ribavirin) within the past 4 weeks before enrollment;
* Subjects who received the live attenuated influenza virus vaccine within the past 21 days;
* Subjects treated with systemic steroids or immunosuppressants within 2 weeks of study start.
* History of alcohol/drug abuse within 6 months of the study start;
* Consumption of >3 alcoholic units for males and females over the past 24 hours. One unit is equivalent to 8 grams of alcohol: a half-pint (~240 milliliter [mL]) of beer; 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period;
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer);
* Exposure to more than four investigational medicinal products within 12 months prior to the first dosing day.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- United States (5):
  - GSK Investigational Site, Palmetto Bay, Florida
  - GSK Investigational Site, Blackfoot, Idaho
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Marshfield, Wisconsin
- Australia (20):
  - GSK Investigational Site, Baulkham Hills, New South Wales
  - GSK Investigational Site, Brookvale, New South Wales
  - GSK Investigational Site, Hinchinbrook, New South Wales
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Browns Plains, Queensland
  - GSK Investigational Site, Everton Plaza, Queensland
  - GSK Investigational Site, Kedron, Queensland
  - GSK Investigational Site, Springfield, Queensland
  - GSK Investigational Site, Glenelg East, South Australia
  - GSK Investigational Site, Happy Valley, South Australia
  - GSK Investigational Site, Berwick, Victoria
  - GSK Investigational Site, Lynbrook, Victoria
  - GSK Investigational Site, Noble Park, Victoria
  - GSK Investigational Site, Pakenham, Victoria
  - GSK Investigational Site, Tarneit, Victoria
  - GSK Investigational Site, Applecross, Western Australia
  - GSK Investigational Site, Baldivis, Western Australia
  - GSK Investigational Site, Claremont, Western Australia
  - GSK Investigational Site, Morley, Western Australia
  - GSK Investigational Site, Yokine, Western Australia
- South Africa (7):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Moloto South, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Western Cape, Western Province
  - GSK Investigational Site, Reiger Park

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=201682

REFERENCES:
- [Background] Roberts G, Chen S, Yates P, Madan A, Walker J, Washburn ML, Peat AJ, Soucie G, Kerwin E, Roy-Ghanta S. Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, and Clinical Effect of Danirixin in Adults With Acute, Uncomplicated Influenza. Open Forum Infect Dis. 2019 Apr 22;6(4):ofz072. doi: 10.1093/ofid/ofz072. eCollection 2019 Apr. PMID 31024969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 45 healthy adult participants with acute, uncomplicated influenza were enrolled. The study was conducted from 01-June 2015 to 25-April-2016 at 17 centres in 3 countries.
Pre-assignment Details: A total of 288 participants were screened for this study. Of these, 243 participants were screen failures and 45 were randomized. The reasons for screen failure included: not meeting inclusion/exclusion criteria (238 participants), lost to follow up (1 participant), investigator discretion (1 participant) and withdrew consent (43 participants).
Groups:
- Danirixin (DNX) 75 mg: Participants received 75 milligram (mg) oral danirixin twice daily with oseltamivir matching placebo twice daily for a total of ten doses over five days
- Placebo (PBO): Participants received danirixin matching placebo twice daily with oseltamivir matching placebo twice daily for a total of ten doses over five days
- Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg: Participants received 75 mg oral danirixin twice daily with 75 mg oseltamivir twice daily for a total of ten doses over five days
- Oseltamivir (OSV) 75 mg: Participants received danirixin matching placebo twice daily with 75 mg oseltamivir twice daily for a total of ten doses over five days
Period: Overall Study
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Started | 15 | 7 | 16 | 7
Completed | 14 | 6 | 14 | 5
Not Completed | 1 | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg | Total
Number analyzed (Participants) | 15 | 7 | 16 | 7 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (13.40) | 33.4 (11.56) | 42.6 (11.53) | 36.3 (9.83) | 38.6 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7 | 2 | 16
  Male | 9 | 6 | 9 | 5 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 2 | 0 | 1 | 1 | 4
  American Indian or Alaskan Native | 1 | 0 | 0 | 0 | 1
  Asian - Central/South Asian Heritage | 0 | 2 | 0 | 0 | 2
  Asian - East Asian Heritage | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 1
  White - White/Caucasian/European Heritage | 11 | 5 | 13 | 6 | 35
  Mixed Race | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to Day 28/withdrawal
Population: Safety population comprised of all randomized participants who received at least one dose of investigational product (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Participants
  AE | 3 | 4 | 7 | 0
  SAE | 1 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Hematology Parameters-Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils (Total Absolute Neutrophil Count [Total ANC]), Platelet Count and White Blood Cell (WBC) Count
Description: Hematology parameters included Basophils, Eosinophils, Lymphocytes, Monocytes, Total neutrophils (Total ANC), Platelet count and WBC count. Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per litre (GI/L)
Groups:
- Danirixin (DNX) 75 Milligram (mg): Participants received 75 mg oral Danirixin twice daily with Oseltamivir matching placebo (PBO [OSV]) twice daily for a total of ten doses over five days
- Placebo (PBO): Participants received Danirixin matching placebo (PBO [DNX]) twice daily with Oseltamivir matching placebo twice daily for a total of ten doses over five days
Arm/Group | Danirixin (DNX) 75 Milligram (mg) | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Giga cells per litre (GI/L)
  Basophils: Day 3: number analyzed (Participants) | 14 | 5 | 12 | 5
  Basophils: Day 3 | -0.011 (0.0511) | -0.002 (0.0377) | -0.008 (0.0196) | -0.008 (0.0130)
  Basophils: Day 5: number analyzed (Participants) | 14 | 6 | 12 | 5
  Basophils: Day 5 | -0.009 (0.0569) | 0.017 (0.0427) | -0.007 (0.0172) | -0.002 (0.0110)
  Basophils: Day 8: number analyzed (Participants) | 14 | 6 | 13 | 5
  Basophils: Day 8 | -0.008 (0.0634) | 0.013 (0.0356) | 0.005 (0.0190) | 0.008 (0.0311)
  Basophils: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 11 | 5
  Basophils: Day 28/withdrawal | -0.007 (0.0517) | 0.003 (0.0287) | 0.030 (0.0520) | 0.010 (0.0332)
  Eosinophils: Day 3: number analyzed (Participants) | 14 | 5 | 12 | 5
  Eosinophils: Day 3 | 0.017 (0.0929) | 0.026 (0.0477) | -0.012 (0.1378) | -0.012 (0.0661)
  Eosinophils: Day 5: number analyzed (Participants) | 14 | 6 | 12 | 5
  Eosinophils: Day 5 | 0.034 (0.1048) | 0.035 (0.0846) | 0.012 (0.1856) | 0.136 (0.3057)
  Eosinophils: Day 8: number analyzed (Participants) | 14 | 6 | 13 | 5
  Eosinophils: Day 8 | 0.074 (0.1248) | 0.078 (0.1332) | 0.036 (0.1416) | -0.000 (0.0959)
  Eosinophils: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 11 | 5
  Eosinophils: Day 28/withdrawal | 0.030 (0.1335) | 0.163 (0.2016) | 0.032 (0.1432) | -0.018 (0.0487)
  Lymphocytes: Day 3: number analyzed (Participants) | 14 | 5 | 12 | 5
  Lymphocytes: Day 3 | 0.093 (0.6701) | 0.778 (0.5904) | 0.463 (0.5443) | 0.432 (0.5124)
  Lymphocytes: Day 5: number analyzed (Participants) | 14 | 6 | 12 | 5
  Lymphocytes: Day 5 | 0.557 (0.7137) | 1.038 (0.7784) | 0.813 (0.6445) | 0.576 (0.3765)
  Lymphocytes: Day 8: number analyzed (Participants) | 14 | 6 | 13 | 5
  Lymphocytes: Day 8 | 0.716 (0.7584) | 1.275 (0.8948) | 0.918 (0.9233) | 0.722 (0.5434)
  Lymphocytes: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 11 | 5
  Lymphocytes: Day 28/withdrawal | 0.564 (0.5969) | 1.619 (0.7884) | 0.903 (0.6779) | 0.788 (0.4467)
  Monocytes: Day 3: number analyzed (Participants) | 14 | 5 | 12 | 5
  Monocytes: Day 3 | -0.117 (0.1524) | -0.178 (0.1970) | -0.105 (0.1927) | -0.070 (0.1562)
  Monocytes: Day 5: number analyzed (Participants) | 14 | 6 | 12 | 5
  Monocytes: Day 5 | -0.175 (0.2817) | -0.128 (0.1631) | -0.090 (0.2479) | -0.118 (0.2104)
  Monocytes: Day 8: number analyzed (Participants) | 14 | 6 | 13 | 5
  Monocytes: Day 8 | -0.104 (0.2310) | -0.097 (0.1425) | -0.108 (0.2043) | 0.024 (0.1730)
  Monocytes: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 11 | 5
  Monocytes: Day 28/withdrawal | -0.061 (0.1785) | -0.011 (0.2230) | -0.016 (0.2232) | 0.064 (0.1343)
  Total neutrophils: Day 3: number analyzed (Participants) | 14 | 5 | 12 | 5
  Total neutrophils: Day 3 | -1.614 (2.1846) | -2.276 (1.5252) | -1.791 (1.9580) | -0.416 (1.0604)
  Total neutrophils: Day 5: number analyzed (Participants) | 14 | 6 | 12 | 5
  Total neutrophils: Day 5 | -1.371 (2.1110) | -1.223 (2.2278) | -0.677 (1.6269) | -0.424 (0.7956)
  Total neutrophils: Day 8: number analyzed (Participants) | 14 | 6 | 13 | 5
  Total neutrophils: Day 8 | 0.463 (2.0336) | -0.830 (2.0826) | -0.137 (2.4279) | 1.766 (2.4391)
  Total neutrophils:Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 11 | 5
  Total neutrophils:Day 28/withdrawal | -0.217 (2.2068) | -0.217 (2.0710) | -0.381 (2.1920) | 0.970 (1.8349)
  Platelet count: Day 3: number analyzed (Participants) | 13 | 6 | 14 | 5
  Platelet count: Day 3 | -9.5 (16.13) | 4.3 (17.68) | -6.1 (17.68) | -3.0 (16.08)
  Platelet count: Day 5: number analyzed (Participants) | 14 | 6 | 14 | 5
  Platelet count: Day 5 | 16.4 (22.92) | 6.7 (21.70) | 13.7 (31.50) | 10.4 (17.78)
  Platelet count: Day 8: number analyzed (Participants) | 14 | 7 | 13 | 5
  Platelet count: Day 8 | 64.3 (45.02) | 62.1 (58.12) | 53.3 (61.73) | 66.2 (22.20)
  Platelet count: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 13 | 5
  Platelet count: Day 28/withdrawal | 28.3 (38.74) | 47.7 (40.13) | 19.2 (42.67) | 44.2 (8.76)
  WBC count: Day 3: number analyzed (Participants) | 14 | 5 | 14 | 5
  WBC count: Day 3 | -1.62 (1.949) | -1.64 (0.879) | -1.49 (1.624) | -0.06 (0.691)
  WBC count: Day 5: number analyzed (Participants) | 14 | 7 | 14 | 5
  WBC count: Day 5 | -0.94 (2.408) | -0.39 (1.676) | -0.17 (1.618) | 0.18 (1.221)
  WBC count: Day 8: number analyzed (Participants) | 14 | 7 | 14 | 5
  WBC count: Day 8 | 1.14 (2.676) | 0.49 (1.842) | 0.79 (2.309) | 2.52 (2.797)
  WBC count: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 13 | 5
  WBC count: Day 28/withdrawal | 0.31 (2.310) | 1.56 (1.992) | 0.51 (2.250) | 1.76 (1.696)

3. Primary Outcome: Change From Baseline in Hematology Parameters- Hemoglobin
Description: Hematology parameters included Hemoglobin. Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Litre (G/L)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Grams per Litre (G/L)
  Day 3: number analyzed (Participants) | 14 | 6 | 14 | 5
  Day 3 | 0.0 (6.08) | 2.2 (5.78) | -4.4 (6.87) | -8.8 (9.78)
  Day 5: number analyzed (Participants) | 14 | 7 | 14 | 5
  Day 5 | -1.3 (6.37) | 0.4 (4.96) | -5.9 (10.87) | -7.4 (11.28)
  Day 8: number analyzed (Participants) | 14 | 7 | 14 | 5
  Day 8 | -5.2 (6.27) | -0.6 (4.65) | -6.1 (11.65) | -7.0 (13.77)
  Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 13 | 5
  Day 28/withdrawal | -5.9 (9.61) | -5.1 (4.49) | -10.1 (7.83) | -4.4 (12.14)

4. Primary Outcome: Change From Baseline in Hematology Parameters- Hematocrit
Description: Hematology parameters included Hematocrit. Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Fraction
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Fraction
  Day 3: number analyzed (Participants) | 14 | 6 | 14 | 5
  Day 3 | -0.0051 (0.01940) | 0.0050 (0.01917) | -0.0126 (0.02310) | -0.0294 (0.03218)
  Day 5: number analyzed (Participants) | 14 | 7 | 14 | 5
  Day 5 | -0.0056 (0.01917) | -0.0029 (0.01734) | -0.0182 (0.03470) | -0.0250 (0.03033)
  Day 8: number analyzed (Participants) | 14 | 7 | 14 | 5
  Day 8 | -0.0173 (0.01958) | -0.0063 (0.01612) | -0.0176 (0.03636) | -0.0244 (0.04140)
  Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 13 | 5
  Day 28/withdrawal | -0.0224 (0.02773) | -0.0171 (0.01933) | -0.0331 (0.02586) | -0.0136 (0.03978)

5. Primary Outcome: Change From Baseline in Hematology Parameters- Mean Corpuscle Hemoglobin (MCH)
Description: Hematology parameters included Mean corpuscle hemoglobin (MCH). Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram (PG)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Picogram (PG)
  Day 3: number analyzed (Participants) | 14 | 6 | 14 | 5
  Day 3 | 0.03 (0.334) | -0.23 (0.242) | -0.21 (0.218) | 0.06 (0.329)
  Day 5: number analyzed (Participants) | 14 | 7 | 14 | 5
  Day 5 | -0.11 (0.407) | -0.19 (0.121) | -0.14 (0.609) | 0.02 (0.455)
  Day 8: number analyzed (Participants) | 14 | 7 | 14 | 5
  Day 8 | -0.16 (0.363) | -0.13 (0.198) | -0.24 (0.477) | 0.08 (0.277)
  Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 13 | 5
  Day 28/withdrawal | 0.12 (0.638) | -0.00 (0.231) | 0.18 (0.479) | 0.20 (0.381)

6. Primary Outcome: Change From Baseline in Hematology Parameters- Mean Corpuscle Volume (MCV)
Description: Hematology parameters included Mean corpuscle volume (MCV). Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters (FL)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Femtoliters (FL)
  Day 3: number analyzed (Participants) | 14 | 6 | 14 | 5
  Day 3 | -0.9 (1.38) | -0.8 (1.17) | -0.4 (1.70) | -0.2 (0.84)
  Day 5: number analyzed (Participants) | 14 | 7 | 14 | 5
  Day 5 | -0.7 (1.20) | -1.3 (1.50) | -0.4 (0.85) | -0.2 (0.84)
  Day 8: number analyzed (Participants) | 14 | 7 | 14 | 5
  Day 8 | -0.6 (1.55) | -1.1 (1.07) | -0.5 (1.02) | -0.4 (1.14)
  Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 13 | 5
  Day 28/withdrawal | -0.4 (2.06) | -0.3 (2.06) | 0.1 (1.04) | 0.6 (0.55)

7. Primary Outcome: Change From Baseline in Hematology Parameters- Red Blood Cell (RBC) Count and Reticulocytes Count
Description: Hematology parameters included RBC count and Reticulocytes count. Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per Liter (TI/L)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Trillion cells per Liter (TI/L)
  RBC: Day 3: number analyzed (Participants) | 14 | 6 | 14 | 5
  RBC: Day 3 | -0.01 (0.209) | 0.13 (0.197) | -0.11 (0.235) | -0.32 (0.370)
  RBC: Day 5: number analyzed (Participants) | 14 | 7 | 14 | 5
  RBC: Day 5 | -0.01 (0.203) | 0.06 (0.190) | -0.19 (0.390) | -0.28 (0.363)
  RBC: Day 8: number analyzed (Participants) | 14 | 7 | 14 | 5
  RBC: Day 8 | -0.13 (0.194) | 0.01 (0.146) | -0.17 (0.389) | -0.28 (0.476)
  RBC: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 13 | 5
  RBC: Day 28/withdrawal | -0.22 (0.272) | -0.16 (0.113) | -0.38 (0.283) | -0.20 (0.464)
  Reticulocytes: Day 3: number analyzed (Participants) | 14 | 6 | 14 | 5
  Reticulocytes: Day 3 | -0.00989 (0.032767) | -0.00392 (0.018792) | -0.01735 (0.025837) | -0.01694 (0.029436)
  Reticulocytes: Day 5: number analyzed (Participants) | 14 | 7 | 14 | 5
  Reticulocytes: Day 5 | -0.01793 (0.023690) | -0.00314 (0.025877) | -0.02635 (0.024815) | -0.01406 (0.024957)
  Reticulocytes: Day 8: number analyzed (Participants) | 14 | 7 | 14 | 5
  Reticulocytes: Day 8 | -0.00158 (0.038763) | -0.00546 (0.022484) | -0.01032 (0.032152) | 0.01020 (0.006260)
  Reticulocytes: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 12 | 5
  Reticulocytes: Day 28/withdrawal | 0.00071 (0.020099) | 0.02313 (0.018277) | -0.00477 (0.030198) | 0.01528 (0.018000)

8. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters- Albumin and Total Protein
Description: Clinical chemistry parameters included Albumin and Total protein. Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Litre (G/L)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Grams per Litre (G/L)
  Albumin: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Albumin: Day 3 | -1.9 (2.12) | -1.7 (2.87) | -2.3 (3.15) | -3.0 (4.42)
  Albumin: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Albumin: Day 5 | -1.8 (1.90) | -1.0 (2.08) | -2.3 (4.37) | -2.6 (1.95)
  Albumin: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Albumin: Day 8 | -1.8 (2.75) | -0.3 (2.50) | -1.7 (4.12) | -0.4 (3.36)
  Albumin: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Albumin: Day 28/withdrawal | -1.6 (2.21) | 0.4 (1.62) | -1.5 (2.24) | 0.2 (3.49)
  Total protein: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Total protein: Day 3 | -1.9 (2.84) | -2.3 (4.61) | -2.8 (4.55) | -4.4 (5.32)
  Total protein: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Total protein: Day 5 | -1.9 (2.20) | -1.3 (3.25) | -2.9 (5.54) | -4.0 (4.06)
  Total protein: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Total protein: Day 8 | -1.3 (2.92) | 0.4 (2.88) | -1.4 (5.77) | -2.2 (5.07)
  Total protein: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Total protein: Day 28/withdrawal | -3.7 (3.41) | -1.0 (2.94) | -3.2 (4.14) | -1.0 (5.24)

9. Primary Outcome: Change From Baseline in Clinical Chemistry- Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST) and Gamma Glutamyl Transferase (GGT)
Description: Clinical chemistry parameters included Alkaline phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase and Gamma Glutamyl Transferase. Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International Units per litre (IU/L)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
International Units per litre (IU/L)
  ALP: Day 3 | -5.0 (6.59) | -5.0 (5.48) | -4.5 (6.52) | -7.2 (9.04)
  ALP: Day 5 | -5.4 (10.96) | -1.9 (6.12) | -4.5 (8.83) | -5.8 (5.26)
  ALP: Day 8 | -4.4 (8.30) | -0.9 (8.32) | 2.9 (9.32) | 0.8 (8.56)
  ALP: Day 28/withdrawal | -2.8 (9.06) | 4.9 (7.43) | -3.8 (7.94) | -1.6 (9.84)
  ALT: Day 3 | 7.9 (28.12) | -0.1 (4.14) | 0.1 (5.25) | -8.4 (8.38)
  ALT: Day 5 | 4.2 (15.27) | 2.4 (7.18) | 0.9 (10.70) | -11.8 (12.50)
  ALT: Day 8 | 2.9 (3.92) | 9.1 (10.98) | 2.7 (15.18) | -11.0 (20.65)
  ALT: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 7
  ALT: Day 28/withdrawal | 2.5 (5.00) | 2.4 (9.69) | -2.9 (11.84) | -12.8 (23.64)
  AST: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  AST: Day 3 | 6.3 (22.53) | 2.9 (5.87) | -0.9 (4.60) | -7.2 (4.49)
  AST: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  AST: Day 5 | 0.9 (4.10) | 2.4 (4.76) | -2.8 (8.33) | -9.4 (5.94)
  AST: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  AST: Day 8 | -0.8 (5.48) | 3.4 (4.54) | -3.3 (7.55) | -10.4 (8.91)
  AST: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  AST: Day 28/withdrawal | -0.2 (6.75) | -1.9 (4.18) | -4.9 (7.62) | -9.8 (11.48)
  GGT: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  GGT: Day 3 | 9.3 (28.87) | 1.0 (4.08) | 0.9 (3.45) | -2.6 (3.13)
  GGT: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  GGT: Day 5 | 7.4 (22.36) | 5.0 (6.58) | 0.8 (5.14) | 0.2 (5.63)
  GGT: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  GGT: Day 8 | 3.3 (11.11) | 7.4 (8.12) | 1.5 (7.50) | 0.2 (10.50)
  GGT: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  GGT: Day 28/withdrawal | -7.6 (17.60) | -1.1 (5.79) | -3.5 (10.62) | -0.6 (15.44)

10. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters- Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid
Description: Clinical chemistry parameters included Direct Bilirubin, Total Bilirubin, Creatinine and Uric acid. Blood samples were collected on Day 1, Day 3, Day 5 and Day28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromole per Liter (UMOL/L)
Groups:
- Danirixin (DNX) 75 Milligram (mg): Participants received 75 milligram (mg) oral danirixin twice daily with oseltamivir matching placebo twice daily for a total of ten doses over five days
Arm/Group | Danirixin (DNX) 75 Milligram (mg) | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Micromole per Liter (UMOL/L)
  Direct Bilirubin: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Direct Bilirubin: Day 3 | -0.3 (0.88) | 0.0 (1.73) | -0.5 (0.74) | 0.2 (0.45)
  Direct Bilirubin: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Direct Bilirubin: Day 5 | -0.5 (0.83) | -0.6 (1.13) | -0.5 (0.74) | 0.2 (0.45)
  Direct Bilirubin: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Direct Bilirubin: Day 8 | 0.1 (0.73) | -0.1 (1.46) | -0.1 (0.83) | 0.0 (1.41)
  Direct Bilirubin:Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Direct Bilirubin:Day 28/withdrawal | 0.1 (1.23) | -0.1 (1.21) | -0.1 (0.83) | 0.0 (0.00)
  Total Bilirubin: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Total Bilirubin: Day 3 | -1.0 (2.30) | -2.0 (7.46) | -1.6 (2.10) | -0.8 (1.79)
  Total Bilirubin: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Total Bilirubin: Day 5 | -1.2 (2.73) | -2.7 (6.37) | 0.0 (2.56) | 1.0 (1.41)
  Total Bilirubin: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Total Bilirubin: Day 8 | -0.9 (1.99) | -0.9 (6.72) | 0.5 (3.09) | 2.2 (3.49)
  Total Bilirubin:Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Total Bilirubin:Day 28/withdrawal | 0.1 (3.45) | -0.3 (6.13) | 0.5 (3.11) | 2.0 (2.45)
  Creatinine: Day 3;: number analyzed (Participants) | 15 | 7 | 15 | 5
  Creatinine: Day 3; | -1.47 (7.891) | -4.39 (6.733) | -6.58 (12.081) | -8.14 (11.291)
  Creatinine: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Creatinine: Day 5 | -4.38 (6.330) | -7.39 (7.240) | -10.16 (14.060) | -11.12 (9.955)
  Creatinine: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Creatinine: Day 8 | -5.79 (7.262) | -10.70 (10.266) | -8.87 (13.815) | -10.32 (5.273)
  Creatinine: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Creatinine: Day 28/withdrawal | -2.54 (5.166) | -4.99 (12.990) | -8.24 (11.771) | -5.34 (5.490)
  Uric acid: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Uric acid: Day 3 | -15.1 (31.18) | -9.9 (42.57) | -15.1 (39.17) | -45.8 (36.03)
  Uric acid: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Uric acid: Day 5 | -18.0 (27.46) | -47.4 (39.09) | -16.3 (45.05) | -54.8 (33.69)
  Uric acid: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Uric acid: Day 8 | 20.8 (48.26) | -14.3 (53.04) | 0.9 (27.41) | -13.0 (69.07)
  Uric acid: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Uric acid: Day 28/withdrawal | 30.1 (47.40) | -0.4 (48.19) | 12.5 (45.09) | 40.6 (63.50)

11. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters- Calcium, Carbon Dioxide (CO2) Content/ Bicarbonate, Glucose, Potassium, Sodium and Urea/Blood Urea Nitrogen (BUN)
Description: Clinical chemistry parameters included Calcium, CO2 content/ Bicarbonate, Glucose, Potassium, Sodium and Urea/(BUN). Blood samples were collected on Day 1, Day 3, Day 5 and Day 28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (MMOL/L)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Millimoles per Liter (MMOL/L)
  Calcium: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Calcium: Day 3 | -0.036 (0.0735) | 0.020 (0.0370) | -0.046 (0.1015) | -0.092 (0.1101)
  Calcium: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Calcium: Day 5 | -0.029 (0.0917) | 0.019 (0.0672) | -0.033 (0.1079) | -0.052 (0.0642)
  Calcium: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Calcium: Day 8 | -0.010 (0.0842) | 0.053 (0.0720) | 0.030 (0.0994) | 0.004 (0.1178)
  Calcium: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Calcium: Day 28/withdrawal | -0.019 (0.1077) | 0.099 (0.0334) | 0.031 (0.0842) | 0.098 (0.1274)
  CO2 / Bicarbonate: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  CO2 / Bicarbonate: Day 3 | 0.1 (2.74) | 0.9 (2.34) | 0.3 (2.50) | -1.8 (2.77)
  CO2 / Bicarbonate: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  CO2 / Bicarbonate: Day 5 | 0.4 (2.35) | 0.9 (1.07) | -0.5 (2.45) | -1.4 (3.21)
  CO2 / Bicarbonate: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  CO2 / Bicarbonate: Day 8 | 0.6 (3.10) | -0.1 (1.95) | 0.4 (2.67) | -0.2 (1.10)
  CO2 / Bicarbonate: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  CO2 / Bicarbonate: Day 28/withdrawal | -0.4 (2.59) | 1.1 (3.13) | -0.5 (2.44) | -1.2 (1.64)
  Glucose: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Glucose: Day 3 | 0.28 (1.084) | 0.23 (1.680) | 0.51 (1.385) | 0.62 (0.782)
  Glucose: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Glucose: Day 5 | 0.13 (1.084) | 0.13 (1.529) | 0.29 (1.904) | 1.30 (2.374)
  Glucose: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Glucose: Day 8 | 0.20 (1.301) | -0.16 (1.042) | -0.13 (1.669) | 0.48 (0.733)
  Glucose: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Glucose: Day 28/withdrawal | 0.27 (1.221) | 0.71 (2.685) | 0.43 (1.909) | 0.22 (0.760)
  Potassium: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Potassium: Day 3 | -0.12 (0.351) | 0.13 (0.411) | 0.01 (0.237) | -0.12 (0.396)
  Potassium: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Potassium: Day 5 | -0.07 (0.401) | 0.16 (0.428) | 0.11 (0.317) | 0.08 (0.572)
  Potassium: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Potassium: Day 8 | 0.08 (0.353) | 0.21 (0.285) | 0.15 (0.223) | 0.02 (0.409)
  Potassium: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Potassium: Day 28/withdrawal | -0.04 (0.455) | 0.07 (0.419) | 0.14 (0.422) | 0.24 (0.635)
  Sodium: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Sodium: Day 3 | 0.5 (1.77) | 0.1 (2.41) | 1.4 (1.64) | 2.0 (1.87)
  Sodium: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Sodium: Day 5 | 0.3 (2.82) | 1.1 (1.86) | 0.7 (2.63) | 1.8 (2.39)
  Sodium: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Sodium: Day 8 | 0.9 (2.64) | 0.3 (1.70) | 1.5 (2.33) | 2.4 (1.67)
  Sodium: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Sodium: Day 28/withdrawal | -0.3 (1.82) | 0.6 (2.99) | 0.6 (2.50) | 1.6 (1.34)
  Urea/BUN: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Urea/BUN: Day 3 | 0.31 (0.956) | -0.31 (0.888) | 0.29 (1.046) | -0.24 (1.328)
  Urea/BUN: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Urea/BUN: Day 5 | 0.47 (0.830) | -0.19 (1.194) | 0.32 (1.197) | -0.88 (1.413)
  Urea/BUN: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Urea/BUN: Day 8 | 0.90 (1.563) | 0.17 (1.081) | 0.82 (1.050) | 0.32 (1.134)
  Urea/BUN: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 14 | 5
  Urea/BUN: Day 28/withdrawal | 0.60 (1.091) | 0.96 (2.082) | 1.19 (0.910) | 0.66 (1.324)

12. Primary Outcome: Change From Baseline in Urinalysis Parameters- Urine pH
Description: Urinalysis parameters included urine pH. pH is calculated on a scale of 0 to 14, such that, the lower the number, more acidic the urine and higher the number, more alkaline the urine with 7 being neutral. Urinalysis was done on Day 1, Day 5 and Day 28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1), Day 5 and Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Points on a scale
  Day 5: number analyzed (Participants) | 14 | 7 | 15 | 5
  Day 5 | 0.00 (0.784) | 0.21 (0.951) | 0.20 (0.592) | 0.40 (0.652)
  Day 28/withdrawal: number analyzed (Participants) | 13 | 7 | 14 | 5
  Day 28/withdrawal | 0.27 (0.633) | 0.14 (0.852) | 0.07 (0.938) | 0.70 (0.570)

13. Primary Outcome: Change From Baseline in Urinalysis Parameters- Urine Specific Gravity
Description: Urinalysis parameter included Urine specific gravity and was measured on Day 1, Day 5 and Day 28. Urinary specific gravity is a measure of the concentration of solutes in the urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1), Day 5 and Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Ratio
  Day 5: number analyzed (Participants) | 14 | 7 | 15 | 5
  Day 5 | -0.0001 (0.00469) | -0.0004 (0.00675) | -0.0038 (0.00731) | -0.0076 (0.00385)
  Day 28/withdrawal: number analyzed (Participants) | 13 | 7 | 14 | 5
  Day 28/withdrawal | -0.0045 (0.00702) | 0.0013 (0.00929) | -0.0021 (0.00855) | -0.0050 (0.00656)

14. Primary Outcome: Number of Participants With Maximum Post-baseline Urine Dipstick Abnormalities- Urine Occult Blood (Dipstick)
Description: The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine occult blood can be read as negative, Trace, 1+, 2+, 3+ and 4+, indicating proportional concentrations in the urine sample. Assessments recorded on Day 1 were considered as Baseline.
Time Frame: Up to Day 28/withdrawal
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 4 | 2 | 4 | 0
Participants
  1+ | 2 | 1 | 1 |
  2+ | 1 | 1 | 1 |
  3+ | 1 | 0 | 0 |
  4+ | 0 | 0 | 2 |

15. Primary Outcome: Number of Participants With Maximum Post-baseline Urine Dipstick Abnormalities- Urine Glucose (Dipstick)
Description: The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine glucose can be read as negative, Trace, 1+ or 1/4 gram per deciliter (G/dL), 2+ OR 1/2 G/dL, 3+ or 1 G/dL and 4+ indicating proportional concentrations in the urine sample. Assessments recorded on Day 1 were considered as Baseline.
Time Frame: Up to Day 28/withdrawal
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 1 | 1 | 1 | 0
Participants
  1+ OR 1/4 G/DL (%) | 0 | 1 | 0 |
  2+ OR 1/2 G/DL (%) | 1 | 0 | 0 |
  3+ OR 1 G/DL (%) | 0 | 0 | 1 |
  4+ | 0 | 0 | 0 |

16. Primary Outcome: Number of Participants With Maximum Post-baseline Urine Dipstick Abnormalities- Urine Protein (Dipstick)
Description: The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine protein can be read as negative, Trace, 1+, 2+, 3+ and 4+, indicating proportional concentrations in the urine sample. Assessments recorded on Day 1 were considered as Baseline.
Time Frame: Up to Day 28/withdrawal
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 3 | 1 | 3 | 1
Participants
  1+ | 3 | 0 | 3 | 1
  2+ | 0 | 0 | 0 | 0
  3+ | 0 | 1 | 0 | 0
  4+ | 0 | 0 | 0 | 0

17. Primary Outcome: Change From Baseline in Vital Signs- Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Vital signs were measured in semi-supine position after 5 minutes rest and included systolic and diastolic blood pressure. Three readings of blood pressure were taken; the first reading was rejected and the second and third readings were averaged to give the measurement to be recorded. Vital signs were obtained on Baseline (Day 1), Day 3, Day 5, Day 8, Day 14 and Day 28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Millimeters of Mercury (mmHg)
  DBP: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  DBP: Day 3 | -2.1 (8.07) | -0.7 (7.97) | -1.1 (9.18) | -4.2 (3.90)
  DBP: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  DBP: Day 5 | 0.3 (6.76) | -1.1 (8.76) | -2.1 (8.53) | -5.2 (6.98)
  DBP: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  DBP: Day 8 | -4.4 (7.13) | -4.6 (10.36) | -2.3 (7.96) | -0.8 (5.07)
  DBP: Day 14: number analyzed (Participants) | 15 | 7 | 15 | 5
  DBP: Day 14 | -4.5 (7.43) | -0.7 (10.63) | 0.8 (9.66) | -7.8 (4.87)
  DBP: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 6
  DBP: Day 28/withdrawal | -4.4 (10.37) | -0.6 (13.82) | -1.1 (8.18) | -3.5 (6.57)
  SBP: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  SBP: Day 3 | -5.73 (13.599) | -5.29 (8.597) | -2.87 (6.802) | -5.00 (5.568)
  SBP: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  SBP: Day 5 | -3.00 (11.802) | -0.71 (4.923) | -1.93 (11.279) | -3.00 (8.456)
  SBP: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  SBP: Day 8 | -5.86 (19.907) | -9.29 (13.889) | -2.60 (13.741) | 0.60 (10.164)
  SBP: Day 14: number analyzed (Participants) | 15 | 7 | 15 | 5
  SBP: Day 14 | -6.20 (12.260) | -4.57 (10.163) | -1.20 (12.667) | -3.80 (7.259)
  SBP: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 6
  SBP: Day 28/withdrawal | -3.36 (16.284) | -0.43 (7.115) | -0.80 (6.982) | -2.83 (7.278)

18. Primary Outcome: Change From Baseline in Vital Signs- Heart Rate (HR)
Description: Vital signs were measured in semi-supine position after 5 minutes rest and included HR. Three readings of pulse rate were taken; the first reading was rejected and the second and third readings were averaged to give the measurement to be recorded. Vital signs were obtained on Day 1, Day 3, Day 5, Day 8, Day 14 and Day 28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Beats per minute
  Heart rate: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Heart rate: Day 3 | 3.93 (10.375) | -8.00 (14.855) | -8.87 (11.637) | -1.20 (16.976)
  Heart rate: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Heart rate: Day 5 | -2.60 (7.385) | -10.29 (21.109) | -9.60 (14.161) | -6.80 (12.637)
  Heart rate: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Heart rate: Day 8 | -2.79 (10.297) | -12.29 (21.422) | -10.87 (14.589) | -0.80 (17.541)
  Heart rate: Day 14: number analyzed (Participants) | 15 | 7 | 15 | 5
  Heart rate: Day 14 | 0.80 (13.165) | -13.43 (14.444) | -8.73 (14.553) | -4.20 (17.584)
  Heart rate: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 6
  Heart rate: Day 28/withdrawal | -6.57 (11.043) | -17.14 (19.912) | -11.80 (15.799) | 0.17 (12.952)

19. Primary Outcome: Change From Baseline in Vital Signs- Respiration Rate (RR)
Description: Vital signs were measured in semi-supine position after 5 minutes rest and included RR. RR was obtained on Day 1, Day 3, Day 5, Day 8, Day 14 and Day 28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Breaths per minute
  RR: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  RR: Day 3 | -0.1 (2.03) | 0.0 (2.00) | -0.5 (2.23) | 1.4 (1.95)
  RR: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  RR: Day 5 | -0.5 (2.10) | 0.0 (1.63) | -0.7 (2.58) | 1.2 (1.10)
  RR: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  RR: Day 8 | -0.3 (2.46) | 0.7 (2.21) | -0.6 (2.38) | 0.6 (1.34)
  RR: Day 14: number analyzed (Participants) | 15 | 7 | 15 | 5
  RR: Day 14 | -0.7 (2.66) | 0.6 (2.23) | -0.3 (2.77) | 0.8 (1.10)
  RR: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 6
  RR: Day 28/withdrawal | -0.4 (2.02) | 0.4 (3.46) | -0.3 (2.97) | 0.8 (2.23)

20. Primary Outcome: Change From Baseline in Vital Signs- Temperature
Description: Vital signs were measured in semi-supine position after 5 minutes rest and included temperature. Oral temperature was obtained on Day 1, Day 3, Day 5, Day 8, Day 14 and Day 28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centigrade
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Centigrade
  Temperature: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  Temperature: Day 3 | -0.20 (1.342) | -1.11 (0.749) | -0.57 (0.884) | -0.08 (0.239)
  Temperature: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  Temperature: Day 5 | -0.75 (1.278) | -1.34 (0.978) | -0.76 (0.766) | -0.14 (0.422)
  Temperature: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  Temperature: Day 8 | -0.46 (0.818) | -1.50 (1.127) | -0.83 (0.786) | -0.16 (0.537)
  Temperature: Day 14: number analyzed (Participants) | 15 | 7 | 15 | 5
  Temperature: Day 14 | -0.73 (1.177) | -1.59 (1.051) | -0.83 (0.970) | -0.28 (0.409)
  Temperature: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 6
  Temperature: Day 28/withdrawal | -0.71 (1.240) | -1.39 (0.958) | -0.71 (0.905) | -0.22 (0.454)

21. Primary Outcome: Change From Baseline in Vital Signs- Percent Oxygen in Blood (POB)
Description: Vital signs were measured in semi-supine position after 5 minutes rest and included POB. POB was obtained on Baseline (Day 1), Day 3, Day 5, Day 8, Day 14 and Day 28/withdrawal. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Percentage (%)
  POB: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  POB: Day 3 | -1.7 (3.97) | 1.1 (1.68) | 0.1 (1.60) | 0.4 (2.61)
  POB: Day 5: number analyzed (Participants) | 15 | 7 | 15 | 5
  POB: Day 5 | -0.7 (1.35) | -0.4 (3.10) | 0.4 (1.76) | 1.0 (2.00)
  POB: Day 8: number analyzed (Participants) | 14 | 7 | 15 | 5
  POB: Day 8 | -0.8 (1.31) | 0.4 (1.62) | -0.1 (2.09) | 0.8 (3.70)
  POB: Day 14: number analyzed (Participants) | 15 | 7 | 15 | 5
  POB: Day 14 | -0.7 (1.71) | 0.9 (3.13) | 0.0 (1.77) | 0.8 (2.39)
  POB: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 6
  POB: Day 28/withdrawal | -1.1 (1.83) | 1.1 (1.86) | 0.2 (1.42) | 1.5 (2.88)

22. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters
Description: 12-lead ECGs were obtained on Day 1, Day 3 and Day28/withdrawal using an ECG machine that automatically calculates and measures RR, PR, QRS, QT, and Corrected QT Interval using Bazette's formula (QTcB) and Corrected QT Interval using Fridericia forumula (QTcF) intervals. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and up to Day 28/withdrawal
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Millisecond (msec)
  RR Interval: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  RR Interval: Day 3 | -5.8 (123.37) | 49.4 (75.29) | 83.0 (144.39) | 39.2 (200.77)
  RR Interval: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 5
  RR Interval: Day 28/withdrawal | 58.2 (94.94) | 76.9 (151.52) | 107.4 (195.56) | 41.2 (103.82)
  QT Interval: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  QT Interval: Day 3 | 3.1 (25.90) | 25.0 (19.86) | 17.7 (28.78) | 30.7 (38.72)
  QT Interval: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 5
  QT Interval: Day 28/withdrawal | 18.9 (19.35) | 35.9 (20.36) | 25.3 (39.96) | 11.1 (16.79)
  QTcF: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  QTcF: Day 3 | 4.5 (21.76) | 18.8 (13.90) | 6.5 (12.89) | 24.6 (13.03)
  QTcF:Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 5
  QTcF:Day 28/withdrawal | 11.0 (14.10) | 24.8 (11.73) | 11.0 (18.07) | 4.3 (5.31)
  QTcB: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  QTcB: Day 3 | 4.1 (25.69) | 14.3 (11.93) | 0.3 (12.63) | 20.9 (8.83)
  QTcB: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 5
  QTcB: Day 28/withdrawal | 6.6 (15.25) | 17.0 (22.12) | 3.5 (14.03) | 0.1 (7.16)
  PR Interval: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  PR Interval: Day 3 | 2.4 (6.47) | -5.4 (20.25) | 0.4 (10.53) | 2.3 (10.52)
  PR Interval: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 5
  PR Interval: Day 28/withdrawal | 3.1 (6.33) | 9.3 (11.87) | 3.0 (13.47) | 2.5 (5.27)
  QRS Duration: Day 3: number analyzed (Participants) | 15 | 7 | 15 | 5
  QRS Duration: Day 3 | 1.5 (4.45) | -5.6 (6.47) | -0.5 (6.14) | 1.9 (8.92)
  QRS Duration: Day 28/withdrawal: number analyzed (Participants) | 14 | 7 | 15 | 5
  QRS Duration: Day 28/withdrawal | -1.3 (5.29) | -5.7 (12.47) | 0.6 (8.77) | 0.3 (4.09)

23. Primary Outcome: Number of Participants With Disease Related Events (DREs) of Interest
Description: Disease-related events of interest included Otitis media, Sinusitis, Bronchitis and Pneumonia and were captured separately from AEs and SAEs. DREs of interest were assessed and recorded by the site on all clinical visit days.
Time Frame: Up to Day 28/withdrawal
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Participants | 2 | 0 | 1 | 0

24. Primary Outcome: Number of Participants With DRE of Interest-associated Antibiotic Use
Description: Use of antibiotics for DREs of interest was monitored. Roxithromycin was used for DRE sinusitis by one participant.
Time Frame: Up to Day 28/withdrawal
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Participants | 0 | 0 | 1 | 0

25. Secondary Outcome: Time to Resolution of Fever Over Time Post Initiation of Treatment
Description: Time to resolution of fever was defined as the time when oral temperature was <= 37.2 degree Celsius (<=99.0 degree Fahrenheit) for at least 24 hours (with one hour window) without having taken any antipyretic medication for at least 4 hours. Temperature was taken orally and recorded in the eDiary, thrice daily from Day 1 to Day 5 (morning, noon, evening) and twice daily (morning, evening) from Day 6 to Day 14 by the participant using a digital thermometer provided by the study. For participants whose fever was not resolved by the Day 14 visit then after Day 14, participants continued to take oral temperature twice daily until temperature <=37.2 degree Celsius or <=99 degree Fahrenheit for 24 hours.
Time Frame: Up to Day 28/withdrawal
Population: Influenza positive population (IPP) comprised of all randomized participants who received at least one dose of IP with proven influenza infection (positive rapid antigen test and positive influenza by quantitative reverse transcription-polymerase chain reaction (qRT-PCR) or culture test at any time point). Participants with fever are analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 7 | 6 | 12 | 5
Hours | 119.833 [15.167 to NA] — Missing Kaplan Meier estimates are due to censoring | 98.092 [46.033 to 129.917] | 54.425 [13.833 to NA] — Missing Kaplan Meier estimates are due to censoring | 76.167 [18.150 to NA] — Missing Kaplan Meier estimates are due to censoring

26. Secondary Outcome: Number of Afebrile Participants Over Time Post Initiation of Treatment
Description: Afebrile participants were defined as participants with oral temperature <=37.2 degree Celsius, <=99.0 degree Fahrenheit over time post initiation of treatment. Temperature was taken orally and recorded in the eDiary, thrice daily from Day 1 to Day 5 (morning, noon, evening) and twice daily (morning, evening) from Day 6 to Day 14 by the participant using a digital thermometer provided by the study. For participants whose fever was not resolved by the Day 14 visit then after Day 14, participants continued to take oral temperature twice daily until temperature <=37.2 degree Celsius or <=99 degree Fahrenheit for 24 hours.
Time Frame: Up to Day 28/withdrawal
Population: IPP population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 7 | 6 | 12 | 5
Participants
  At 0 hour | 0 | 0 | 0 | 0
  At 24 hours | 1 | 0 | 2 | 1
  At 72 hours | 2 | 2 | 8 | 2
  At 120 hours | 4 | 4 | 10 | 3
  At 192 hours | 4 | 6 | 11 | 3
  At 336 hours | 5 | 6 | 11 | 3
  At 672 hours | 5 | 6 | 11 | 3

27. Secondary Outcome: Number of Participants Who Used Relief Medication
Description: Use of study supplied relief medications (paracetamol and dextromethorphan for symptom relief were recorded in the eDiary and accordingly number of participants using these medications were recorded.
Time Frame: Up to Day 28/withdrawal
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Participants
  Paracetamol use | 12 | 7 | 15 | 7
  Dextromethorphan use | 12 | 5 | 13 | 7

28. Secondary Outcome: Number of Hospital Admissions Due to Influenza Infection
Description: Number of participants admitted in hospital due to influenza infection was recorded.
Time Frame: Up to Day 28/withdrawal
Population: Safety population
Measure: Number; unit: Participants
Groups:
- Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg; Oseltamivir (OSV) 75 mg: Participants received danirixin matching placebo twice daily with 75 mg oseltamivir twice daily for a total of ten doses over five days
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Participants | 0 | 0 | 0 | 0

29. Secondary Outcome: Change From Baseline in Influenza Viral Load as Measured by Quantitative Reverse Transcription-polymerase Chain Reaction (qRT-PCR) From Nasopharyngeal Swabs on Day 3, Day 5, Day 8 and Day 14
Description: Influenza viral load as measured by quantitative reverse transcription - polymerase chain reaction (qRT-PCR) from nasopharyngeal swabs on Baseline (Day 1), Day 3, Day 5, Day 8 and Day 14 was recorded. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and Day 3, Day 5, Day 8 and Day 14
Population: IPP population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log viral particles/mL
Groups:
- Danirixin (DNX) 75 mg; Placebo (PBO): Participants received danirixin matching placebo twice daily with oseltamivir matching placebo twice daily for a total of ten doses over five days
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 9 | 6 | 13 | 7
Log viral particles/mL
  Day 3: number analyzed (Participants) | 9 | 6 | 12 | 5
  Day 3 | -0.897 (1.1390) | -1.415 (1.5986) | -1.620 (1.3461) | -1.904 (1.6289)
  Day 5: number analyzed (Participants) | 9 | 6 | 12 | 5
  Day 5 | -1.912 (1.2895) | -2.812 (1.8841) | -2.962 (1.8515) | -2.644 (0.5206)
  Day 8: number analyzed (Participants) | 8 | 6 | 12 | 5
  Day 8 | -3.764 (1.8831) | -4.063 (1.4120) | -3.862 (1.3284) | -4.250 (1.7995)
  Day 14: number analyzed (Participants) | 9 | 5 | 12 | 5
  Day 14 | -4.024 (1.0387) | -4.992 (1.1296) | -4.518 (1.2408) | -4.250 (1.7995)

30. Secondary Outcome: Number of Participants With no Detectable Influenza Viral RNA by qRT-PCR From Nasopharyngeal Swabs on Baseline (Day 1), Day 3, Day 5, Day 8 and Day 14
Description: Number of participants with no detectable influenza viral ribonucleic acid (RNA) by qRT-PCR from nasopharyngeal swabs on Baseline (Day1), Day 3, Day 5, Day 8 and Day 14 were recorded. Assessments recorded on Day 1 were considered as Baseline.
Time Frame: Up to Day 14
Population: IPP Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 mg | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 9 | 6 | 13 | 7
Participants
  Day 1 | 0 | 0 | 0 | 0
  Day 3: number analyzed (Participants) | 9 | 6 | 12 | 5
  Day 3 | 0 | 0 | 0 | 0
  Day 5: number analyzed (Participants) | 9 | 6 | 12 | 5
  Day 5 | 0 | 0 | 3 | 1
  Day 8: number analyzed (Participants) | 8 | 6 | 12 | 5
  Day 8 | 3 | 1 | 6 | 5
  Day 14: number analyzed (Participants) | 9 | 5 | 12 | 5
  Day 14 | 5 | 4 | 11 | 5

31. Secondary Outcome: Total Dose of Relief Medication
Description: Use of study supplied relief medications (paracetamol and dextromethorphan for symptom relief were recorded in the eDiary and accordingly number of participants using these medications were recorded. The total dose of these relief medications used by these participants are presented.
Time Frame: Up to Day 28/withdrawal
Population: Safety population. Only those participants using relief medication were analyzed.
Measure: Median (Full Range); unit: Milligrams
Arm/Group | Danirixin (DNX) 75 Milligram (mg) | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 15 | 7 | 16 | 7
Milligrams
  Paracetamol total dose: number analyzed (Participants) | 12 | 7 | 15 | 7
  Paracetamol total dose | 5000.00 [1000.0 to 14000.0] | 9000.00 [500.0 to 71000.0] | 5500.00 [500.0 to 20000.0] | 3000.00 [1000.0 to 12000.0]
  Dextromethorphan total dose: number analyzed (Participants) | 12 | 5 | 13 | 7
  Dextromethorphan total dose | 150.00 [15.0 to 360.0] | 390.00 [120.0 to 2250.0] | 120.00 [30.0 to 2250.0] | 60.00 [15.0 to 300.0]

32. Secondary Outcome: Change From Baseline in Influenza Viral Load as Measured by Quantitative Virus Culture From Nasopharyngeal Swabs on Day 3, Day 5, Day 8 and Day 14
Description: Influenza viral load as measured by quantitative virus culture from nasopharyngeal swabs on Baseline (Day 1), Day 3, Day 5, Day 8 and Day 14 was recorded. Assessments recorded on Day 1 were considered as Baseline. Change from Baseline was equal to Post-Dose Visit Value minus Baseline.
Time Frame: Baseline (Day 1) and Day 3, Day 5, Day 8 and Day 14
Population: IPP population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log median tissue culture infective dose
Arm/Group | Danirixin (DNX) 75 Milligram (mg) | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 9 | 6 | 13 | 7
Log median tissue culture infective dose
  Day 3: number analyzed (Participants) | 9 | 6 | 12 | 5
  Day 3 | -1.810 (1.4374) | -0.753 (1.8251) | -1.943 (2.0079) | -2.304 (1.9351)
  Day 5: number analyzed (Participants) | 9 | 6 | 12 | 5
  Day 5 | -2.534 (1.4499) | -2.172 (1.9242) | -2.467 (1.8842) | -3.108 (2.0998)
  Day 8: number analyzed (Participants) | 8 | 6 | 12 | 5
  Day 8 | -2.885 (1.1877) | -2.843 (2.2061) | -2.698 (1.4621) | -3.108 (2.0998)
  Day 14: number analyzed (Participants) | 9 | 5 | 12 | 5
  Day 14 | -2.564 (1.4694) | -2.260 (1.8792) | -2.614 (1.5899) | -3.108 (2.0998)

33. Secondary Outcome: Number of Participants With no Detectable Influenza Viral RNA by Quantitative Virus Culture From Nasopharyngeal Swabs on Baseline (Day 1), Day 3, Day 5, Day 8 and Day 14
Description: Number of participants with no detectable influenza viral RNA by quantitative virus culture from nasopharyngeal swabs on Baseline (Day1), Day 3, Day 5, Day 8 and Day 14 were recorded. Assessments recorded on Day 1 were considered as Baseline.
Time Frame: Up to Day 14
Population: IPP Population. Only those participants (number with nasopharyngeal samples) available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Danirixin (DNX) 75 Milligram (mg) | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
Number analyzed (Participants) | 9 | 6 | 13 | 7
Participants
  Day 1 | 1 | 0 | 0 | 2
  Day 3: number analyzed (Participants) | 9 | 6 | 12 | 5
  Day 3 | 5 | 2 | 6 | 3
  Day 5: number analyzed (Participants) | 9 | 6 | 12 | 5
  Day 5 | 7 | 3 | 10 | 5
  Day 8: number analyzed (Participants) | 8 | 6 | 12 | 5
  Day 8 | 8 | 6 | 12 | 5
  Day 14: number analyzed (Participants) | 9 | 5 | 12 | 5
  Day 14 | 9 | 5 | 12 | 5

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Safety population comprised of all randomized participants who received at least one dose of investigational product.
Arm/Group | Danirixin (DNX) 75 Milligram (mg) | Placebo (PBO) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg | Oseltamivir (OSV) 75 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7 | 0/16 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/7 | 0/16 | 0/7
Other Adverse Events (participants affected / at risk) | 1/15 | 2/7 | 3/16 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danirixin (DNX) 75 Milligram (mg) (N=15) | Placebo (PBO) (N=7) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg (N=16) | Oseltamivir (OSV) 75 mg (N=7)
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Danirixin (DNX) 75 Milligram (mg) (N=15) | Placebo (PBO) (N=7) | Danirixin (DNX) 75 mg + Oseltamivir (OSV) 75 mg (N=16) | Oseltamivir (OSV) 75 mg (N=7)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.